CLINICAL TRIAL: NCT03146715
Title: The Effect of a Nutrient Dense Food on the Skin Carotenoid Levels of School Age Children
Brief Title: The Effect of a Nutrient Dense Food on the Skin CarotenoidLevels of School Age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: Utah Agriculture Experiment Station (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: USU #6351
Record Dates: First submitted 2017-04-20; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Raman Spectroscopy; Children, Only

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-carotenoid food feeding trial (Active Comparator): Twenty-three children were randomly assigned to a treatment with a high carotenoid baked food (4.3mg carotenoids/120g, 360 kcal)
  Interventions: Other: Feeding trial
- No-carotenoid food feeding trial (Placebo Comparator): Twenty-five children were randomly assigned to consume a baked food with no carotenoids (300 kcals/73g)
  Interventions: Other: Feeding trial

INTERVENTIONS:
Other: Feeding trial — Children were asked to eat the designated portion of the assigned food once a day for six weeks.

SUMMARY:
Background: In a previous study, children who consumed a high-carotenoid juice over 8 weeks significantly increased skin carotenoid levels as compared to children who consumed a placebo juice. A naturally carotenoid-rich baked product, potentially marketable as a healthy breakfast food alternative, was developed by Utah State University researchers.

Objective: To determine the effect and response of a carotenoid-rich baked product on change in skin carotenoid levels among children.

Design: A six week randomized controlled trial. Participants/setting: Participants were children age 5-18 during March-June, 2015 living in Cache County, UT (n=46). Intervention: Children were randomly assigned to one of two groups: treatment (n=23) with a high carotenoid baked food or control (n=25) who consumed a baked food with no carotenoids. Children were asked to eat the designated portion of the assigned food once a day for six weeks. Skin carotenoid levels were measured every two weeks by a BioPhotonic scanner and reported in Raman intensity counts. Participants were asked to maintain their diet and completed a food frequency questionnaire at Baseline, Week 3, and Week 6. Uneaten portions of the food were returned to clinic, counted, and recorded.

Main outcome measures: Change in skin carotenoid levels as measured in Raman counts over 6 weeks.

Statistical analysis performed: Repeated-measures ANOVA was used to assess the group differences in Raman counts.

ELIGIBILITY:
Inclusion Criteria:

* Skin carotenoid levels 11,000-33,000 Raman intensity counts
* Age 5-18 years
* Willing to attend 7 clinic visits
* Willing to eat designated food each day for 6 weeks

Exclusion Criteria:

* Illness in two weeks before study began
* Chronic disease such as asthma, rheumatoid arthritis, type 1 diabetes
* Skin carotenoid levels <11,000 and >33,000 Raman intensity counts
* Consumption of high carotenoid supplements
* Use of topical self-tanning lotion

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Raman resonance spectroscopy | 6 weeks
  The skin carotenoid levels were determined by calculating the average height of the peak Raman absorbance signal obtained and quantified from excitation of skin carotenoids using a low-intensity blue light-emitting diodes light (λ=473 nm) with green light (510 nm) detection.24 The BioPhotonic Scanner Everest 2TM skin carotenoids were reported as Raman intensity counts. The higher the count, the higher the concentration of carotenoid molecules detected at the site of measurement. The scanner reports total carotenoid count, rather than individual carotenoid counts, as there is overlap in the absorption spectra of each carotenoid. During the warm-up process, the black calibration cap, which covers the scanner's light-emitting diodes light, allows the scanner to self-calibrate using a patented process.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Allen, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Center for Human Nutrition Studies, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No